CLINICAL TRIAL: NCT00808951
Title: In Vivo and in Vitro Efficacy of the Recommended First Line Antimalarial Treatments (Artemether-Lumefantrine and Amodiaquine-Artesunate) in Children With Uncomplicated Malaria in Burkina Faso
Brief Title: In Vivo and in Vitro Efficacy of Antimalarial Treatments in Children in Burkina Faso
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Muraz (Other)
Collaborators: Institute of Tropical Medicine, Belgium (Other)
Responsible Party: Principal Investigator, Tinto Halidou, PharmD, PhD, Centre Muraz
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Malactres-BF
Record Dates: First submitted 2008-12-05; First posted 2008-12-16 (Estimated); Last update posted 2015-08-03 (Estimated); Status verified 2015-07

CONDITIONS: Malaria
Keywords: Uncomplicated malaria; P falciparum; Children; National treatment protocol; Burkina Faso; Artemether-lumefantrine; Artesunate-amodiaquine; In vivo efficacy; In vitro efficacy
MeSH Terms: conditions — Malaria | interventions — amodiaquine, artesunate drug combination; Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Artemether -lumefantrine (Experimental): Treatment of malaria with Artemether-lumefantrine (AL), according to one of the two options given by national protocol in Burkina Faso
  Interventions: Drug: Artemether-lumefantrine
- Artesunate-amodiaquine (Experimental): Treatment of malaria with Artesunate-amodiaquine(AS-AQ), according to one of the two options given by national protocol in Burkina Faso
  Interventions: Drug: Artesunate-amodiaquine

INTERVENTIONS:
Drug: Artesunate-amodiaquine — Coformulated AQ+AS by Sanofi-Aventis has been pre-qualified by WHO in 2008. It is administered once daily for three consecutive days, and it is available in three different dosages (25mg/67.5mg; 50mg/135mg; 100mg/270mg)
  Other Names: ASAQ, Coarsucam
  Arms: Artesunate-amodiaquine
Drug: Artemether-lumefantrine — Artemether-lumefantrine by Novartis was the first fixed-dose ACT that was prequalified by WHO in April 2004. A 3-day, 6-dose regimen of AL is recommended for infants and children weighing 5-35 kg and adults weighing > 35 kg.
  Other Names: AL, Coartem(R), Riamet(R)
  Arms: Artemether -lumefantrine

SUMMARY:
Resistance to antimalarial drugs represents a major obstacle for controlling malaria in endemic countries, so that most sub-Saharan countries have changed their antimalarial drug policy to the new Artemisinin Containing Therapies. Burkina Faso has changed its policy for uncomplicated malaria to Artemether-Lumefantrine (AL) and Artesunate-Amodiaquine (AQ+AS), but there are still little available data on safety and efficacy of these treatments in Burkina Faso; both treatments have shown to be efficacious, but AL seems to have higher occurrence of recurrent malaria infections during a 28-day follow up period. Thus, this study aims at comparing the safety and efficacy of AL and AS-AQ (42-day follow-up), AND also at comparing their in vitro sensitivity, in patients with recurrent infection, with the results obtained in vivo.

DETAILED DESCRIPTION:
Plasmodium falciparum resistance to antimalarial drugs represents the major drawback and obstacle for controlling malaria in endemic countries; that's why most sub-Saharan countries have changed their antimalarial drug policy to Artemisinin Containing Therapies (ACT), which produce a rapid clinical and parasitological cure, reduce gametocyte carriage rate and are generally well tolerated. Burkina Faso has recently changed its policy for the treatment of uncomplicated malaria, from Chloroquine to Artemether-Lumefantrine (AL) and Artesunate-Amodiaquine (AQ+AS). However, there are still little available data on safety and efficacy of these treatments in Burkina Faso; a recent study carried out in Bobo Dioulasso showed that both treatments were extremely efficacious (adjusted treatment failure less than 5%) but with AL showing significantly high occurrence of recurrent infections during the 28-day follow up period. The higher risk for recurrent infections for AL was confirmed in a subsequent trial comparing AL with AQ-SP and dihydroartemisinin-piperaquine, but so far no direct comparison between AQ+AS and AL has been completed, though a study in Nanoro, near Ouagadougou, is ongoing. Thus, the present study aims at comparing the in vivo safety and efficacy of AL and AS-AQ (42-day follow-up),AND at comparing the in vitro sensitivity of the different ACT components, in patients with recurrent infection, with the results obtained in vivo.

ELIGIBILITY:
Inclusion Criteria:

* Age 6 - 59 months
* Weight > 5 kg
* Mono-infection with P. falciparum
* Parasitemia of 4,000-200,000 asexual parasites per µl
* Fever: > 37.5 °C or history of fever in the preceding 24 hours
* Haemoglobin > 5.0 g/dl
* Signed informed consent by the parents or guardians
* Parents' or guardians' willingness and ability to comply with the study protocol for the duration of the trial.

Exclusion Criteria:

* Participation in any other clinical trial during the previous 30 days
* Known hypersensitivity to the study drugs
* Severe and/or complicated malaria (cases will be referred to Bobo-Dioulasso University hospital for treatment)
* Danger signs: not able to drink or breast-feed, vomiting (> twice in 24hours), recent history of convulsions (>1 in 24h), unconscious state, unable to sit or stand;
* Known intercurrent illness or any condition which would place the subject at undue risk or interfere with the results of the study.
* Severe malnutrition (weight for height <70% of the median NCHS/WHO reference)

Ages: 6 Months to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 440 (Actual)
Dates: Start 2008-12; Primary Completion 2010-10 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
PCR unadjusted treatment failure (regardless of genotyping). | 42 days

SECONDARY OUTCOMES:
PCR adjusted treatment failure | 42 days
PCR unadjusted treatment failure | 28 days
PCR adjusted treatment failure | 28 days
Fever clearance time | day 1, 2, 3
Asexual parasite clearance time | day 7, 14, 21, 28, 35, 42
Gametocytaemia (prevalence and density) | Day 7, 14, 21, 28, 35 and 42
Safety profiles of the two treatments | 42 days overall
Parasites in vitro sensitivity to the drugs tested and their relationship with the in vivo results | before treatment and at the day of reccurrente parasitemia

CONTACTS AND LOCATIONS:
Overall Officials: Halidou Tinto, PhD, Principal Investigator — Centre Muraz
Locations (1):
- Tinto Halidou, Bobo-Dioulasso, Houet, Burkina Faso

REFERENCES:
- [Derived] Lingani M, Bonkian LN, Yerbanga I, Kazienga A, Valea I, Sorgho H, Ouedraogo JB, Mens PF, Schallig HDFH, Ravinetto R, d'Alessandro U, Tinto H. In vivo/ex vivo efficacy of artemether-lumefantrine and artesunate-amodiaquine as first-line treatment for uncomplicated falciparum malaria in children: an open label randomized controlled trial in Burkina Faso. Malar J. 2020 Jan 6;19(1):8. doi: 10.1186/s12936-019-3089-z. PMID 31906948